CLINICAL TRIAL: NCT03383952
Title: A Phase I Trial of CD19 Targeted ICAR19 T Cells in Patients With CD19+ Leukemia and Lymphoma.
Brief Title: A Clinical Study of CD19 Targeted CAR-T for Patients With CD19+ Lymphoma and Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immune Cell, Inc. (Industry)
Collaborators: Weifang People's Hospital (Other)
Responsible Party: Principal Investigator, Xiulian Sun, Principal Investigator, Immune Cell, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19 Targeted CAR-T
Record Dates: First submitted 2017-12-06; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: B Cell Leukemia; B Cell Lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell | interventions — Biological Products

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICAR19 CAR-T cells (Experimental): Immunotherapy offers an extremely precise approach with the potential to eliminate cancer cells specifically. The newly designed CD19 targeted ICAR19 T cells can specifically kill CD19+ tumor cells. ICAR19 CART used the second generation of CART designation. In this study, the participants will receive several doses of autologous ICAR19 CAR-T cells and the investigators will determine the safety and therapeutic effects of these cells.
  Interventions: Biological: ICAR19 CAR-T cells

INTERVENTIONS:
Biological: ICAR19 CAR-T cells — T cells were isolated from peripheral blood from patients enrolled. T cells were transduced with lentivirus bearing anti-CD19 antibody scFV and the activation signals of second generation CART designation. The CART cells were infused into the patients by IV with an escalating dosage.
  Other Names: Biological drug

SUMMARY:
Immunotherapy offers an extremely precise approach with the potential to eliminate cancer cells specifically. The newly designed CD19 targeted ICAR19 T cells can specifically kill CD19+ tumor cells. ICAR19 CART used the second generation of CART designation. In this study, the participants will receive several doses of autologous ICAR19 T cells and the investigators will determine the safety and therapeutic effects of these cells.

ELIGIBILITY:
Inclusion Criteria:

CD19 positive leukemia and lymphoma，relapsed and/or refractory：

* survival>12 weeks;
* FEV1, FVC and DLCO ≥50% of expected corrected for hemoglobin;
* LVEF≥50%;
* Creatinine<2.5mg/dl;
* Bilirubin<2.5mg/dl;
* ALT (alanine aminotransferase)/AST (aspartate aminotransferase)<3 x normal;
* At least 7 days after last chemotherapy;
* provide with informed consent.

Exclusion Criteria:

* Active clinically significant CNS dysfunction
* Pregnant or breast-feeding women.
* Uncontrolled active infection including hepatitis B or C.
* HIV positive.
* Use of systemic steroids within 72 hours.
* Allogeneic lymphocyte treatments within recent 6 months.
* Any uncontrolled active medical disorder.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the safety of ICAR19 CAR-T cells | 2 years
  To assess the adverse events of ICAR19 T cells infusion in patients with CD19+ malignancies

SECONDARY OUTCOMES:
Measure the anti-tumor effect of ICAR19 CAR-T cells | 3 years
  Assess for the therapeutic effects of ICAR 19 CAR-T cells in CD19-expressing leukemia and lymphoma
Survival time of ICAR19 T cells in vivo. | 5 years
  To measure the survival time of ICAR19 CAR-T cells in vivo, extra blood will be drawn from patients receive ICAR19 T cells infusion in the follow-up time

CONTACTS AND LOCATIONS:
Locations (1):
- Weifang People's Hospital, Weifang, Shandong, China